CLINICAL TRIAL: NCT05400252
Title: Whole Health in VA Mental Health: A Randomized Controlled Trial of Omnis Salutis
Brief Title: Whole Health in VA Mental Health: Omnis Salutis
Acronym: OS RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: D3938-R; 1I01RX003938-01A1 (NIH)
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Stress Disorders, Post-Traumatic; Depressive Disorder; Anxiety Disorders; Substance-Related Disorders
Keywords: Patient Participation; Psychosocial Functioning; Communication; Patient Satisfaction; Patient Preference
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder; Anxiety Disorders; Substance-Related Disorders; Patient Participation; Communication; Patient Satisfaction; Patient Preference | interventions — Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind to participant intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omnis Salutis (Experimental): Omnis Salutis is a Veteran-targeted, Whole Health program for mental health care settings and teaches Veterans the skills to identify and communicate their Whole Health goals to providers and social supports
  Interventions: Behavioral: Omnis Salutis
- Health and Wellness (Active Comparator): Health & Wellness is an educational wellness intervention
  Interventions: Behavioral: Health and Wellness

INTERVENTIONS:
Behavioral: Omnis Salutis — Omnis Salutis is a Veteran-targeted, Whole Health program for mental health care settings and teaches Veterans the skills to identify and communicate their Whole Health goals to providers and social supports
  Arms: Omnis Salutis
Behavioral: Health and Wellness — Health & Wellness is an educational wellness intervention
  Arms: Health and Wellness

SUMMARY:
Recent Veterans of the Afghanistan and Iraq conflicts are presenting in VA care with high rates of posttraumatic stress disorder (PTSD), depression, anxiety, and substance use disorders. Difficulties with social relationships and community reintegration are common functional impairments with these disorders. VA is transforming to a Whole Health, patient-centered system of care that will address these issues as part of health care. In a previous study, Omnis Salutis (OS) was developed with Veteran and clinician input. OS is a three-session intervention in which Veterans learn about Whole Health and practice communicating their health mission to providers and social supports. OS was shown feasible to deliver, acceptable to Veterans, and preliminarily effective at improving physical, mental, and social functioning. This study will use a large, multisite randomized controlled trial to test the impact of OS on Veterans' social and physical functioning and Veteran engagement in mental health care. Results will support broad delivery of OS throughout the VA.

DETAILED DESCRIPTION:
Anticipated Impacts on Veteran Healthcare: Recent Veterans of the Operation Enduring Freedom, Operation Iraqi Freedom and Operation New Dawn (OIF/OEF/OND) conflicts are presenting in VA care with high rates of stress related mental health disorders (posttraumatic stress disorder, depression, anxiety, and alcohol abuse), and reporting significant difficulties with social relationships and community reintegration. Surveys of recent Veterans show that Veterans want the VA to provide mental health care tailored to their concerns and reintegration priorities; while simultaneously, the VA has committed to transforming to a Whole Health patient-centered, system of care. Within this context, Omnis Salutis, a brief, Veteran-focused, Whole Health activation intervention, was developed with a stakeholder advisory panel of Veterans, clinicians, and researchers. Preliminary findings indicate that participation in Omnis Salutis was associated with improvements in physical, mental and social functioning among recent Veterans with stress related mental health disorders.

Project Background: The term "recent Veterans" refers to Veterans who served in the OIF/OEF/OND military operations. Almost 60% (708,062) of recent Veterans who received VA care have been diagnosed with a mental health disorder, most commonly post-traumatic stress disorder (56%), depressive disorders (45%), anxiety disorders (44%), and substance use disorders (21%). Recent Veterans with stress-related mental health disorders experience impairment in functional domains of health (overcoming and managing disease), purpose (meaningful daily activities and participation in society), and community (positive relationships and social networks). Omnis Salutis is a three-session intervention in which Veterans learn about Whole Health and complete a brief Personal Health Inventory, practice creating and delivering MY MAP (Mission/Aspiration/Purpose) to communicate their health mission consistently to their providers and social supports; and identify both formal and informal healing relationships that support their health mission. Omnis Salutis was shown to be acceptable to and feasible in a previous small randomized controlled trial (n = 48). Additionally, analyses of the relationship between participation in Omnis Salutis and outcomes on the Veterans RAND 36-Item Health Survey found a large effect for Bodily Pain improvement, medium effect size for Social Functioning, small effect sizes for Physical Functioning, Emotional Well-Being, Energy/Fatigue, Role Limitations due to Emotional Problems, and General Health. These results are very promising and support further testing of Omnis Salutis.

Project Objectives: The proposed research will test the efficacy of Omnis Salutis, a brief, Veteran-focused, Whole Health activation intervention, in a randomized controlled trial (n = 238). The primary aim of the study is to evaluate the efficacy of Omnis Salutis for improving the physical and social functioning of recent Veterans with stress-related disorders. The secondary aim is to evaluate the efficacy of Omnis Salutis for increasing Veteran engagement in care for stress-related disorders. There is an exploratory aim to Evaluate the processes that underlie the relationship between engagement in care and functioning. This study will provide support for Omnis Salutis as an evidence-based practice and for broader dissemination.

Project Methods: The investigators propose a randomized controlled trial in a sample of 238 Veterans with stress-related mental health disorders recruited from four VA medical centers in Maryland, Washington DC, and West Virginia. Veterans will be randomly assigned to receive three sessions of Omnis Salutis or three sessions of an active control, health, and wellness intervention. Both conditions will be delivered via as VA Video Connect (VVC) telehealth platform or telephone. Participants will complete assessments at baseline, 3-month follow-up, 6-month follow-up, and 12-month follow-up timepoints. Analyses will examine differences in change over time between the two intervention conditions.

ELIGIBILITY:
Inclusion Criteria:

Per medical record review:

* military service since 2001
* Veteran accessed MHC service at designated study site for the first time in the last 6 months OR the first time in the last 6 months after at least a one year gap in mental health care
* have a current diagnosis of:

  * PTSD (309.81)
  * major depressive disorder (296.20-296.23, 296.30-296.33)
  * social anxiety disorder (300.23)
  * panic disorder (300.01)
  * generalized anxiety disorder (300.02)
  * other specified or unspecified anxiety disorder (300.09, 300.00)
  * substance use disorders (303.90, 304.00, 304.10, 304.30)

Exclusion Criteria:

* Per medical record review, current diagnosis of a psychotic disorder meeting criteria established by the VA Serious Mental Illness Treatment, Research, and Evaluation Center (SMITREC):

  * schizophrenic disorders (295.0-295.9)
  * affective psychoses (296.0-296.1, 296.4-296.8)
  * major depression with psychotic features (296.24, 296.34)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Veterans RAND 36-Item Health Survey - Physical Component Summary | 6 months
  overall physical functioning; Item response scales differ but are scored on a 3-, 5-, or 6-point scale (possible range 0-64). Item responses are summed with higher scores indicating better functioning.
Veterans RAND 36-Item Health Survey - Social Functioning Scale | 6 months
  overall social functioning in life; Item response are scored on a 5-point scale (possible range 0-4) with higher scores indicating better functioning.

SECONDARY OUTCOMES:
Altarum Consumer Engagement - Commitment and Navigation subscales | 12 months
  patient engagement in health and healthcare decisions; Item responses are scored on a 5-point scale (possible range 0-4) with higher scores indicating better engagement
VA service use | 12 months
  VA service use data as collected from the electronic medical record

CONTACTS AND LOCATIONS:
Overall Officials: Diana P Whitham, PhD MPH RD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (2):
- United States (2):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No